CLINICAL TRIAL: NCT01058577
Title: A Single Center, Open Study to Evaluate Changes in Serum Electrolytes at Different Glucose Concentrations and Their Impact on a Non-invasive Glucose Monitoring Method
Brief Title: Changes in Serum Electrolytes at Different Glucose Concentrations + Impact on a Non-invasive Glucose Monitoring Method
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Profil Institut für Stoffwechselforschung GmbH (Industry)
Collaborators: Pendragon Medical AG Switzerland (Unknown)
Responsible Party: Christoph Kapitza, MD, Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B1-2001-01
Record Dates: First submitted 2010-01-27; First posted 2010-01-28 (Estimated); Last update posted 2010-01-28 (Estimated); Status verified 2010-01

CONDITIONS: Diabetes Mellitus
Keywords: diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Somatostatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Non-invasive CGMS — A non-invasive continuous glucose monitoring device measured was applied at the wrist and measured skin glucose as an indirect measure of blood glucose every 10 min.
  Other Names: PendraWatch
Procedure: Hyperglycemic glucose clamp — The automated glucose clamp technique was used to control glucose levels at baseline glycemia for 1h, hyperglycemia (16.7 mmol/L) for at least 2.5h and euglycemia (5 mmol/L) for another 2.5h. A continuous somatostatin infusion was initiated after 1h to suppress endogenous insulin secretion. A glucose solution was infused to increase the blood glucose towards the hyperglycemic target level. At approximately t=3.5h the somatostatin infusion was stopped and blood glucose was controlled at the euglycemic target level.
  Other Names: Biostator; Somatostatin

SUMMARY:
In healthy subjects: Continuous monitoring of the glucose concentration in the skin by means of a non-invasive glucose sensor during a glucose clamp when systematically changing the blood glucose concentration (e.g. to hyperglycemia). Simultaneous frequent determinations of serum electrolytes.

DETAILED DESCRIPTION:
Non-invasive continuous glucose monitoring is a promising approach in diabetes therapy. It is known that changes in glucose concentration in the skin can be registered by means of optical, spectroscopic measures in subjects with diabetes. The precision of such measures, however, so far has been unsatisfactory.

This study evaluates the changes in skin glucose concentration by means of a non-invasive glucose sensor and compares these to blood glucose concentrations during a glucose clamp. It is also known that with hyperglycemic blood glucose concentrations there is a consecutive hyponatraemia. This study shall evaluate to which extent and how fast serum electrolyte parameters change when establishing a hyperglycaemic blood glucose level. This shall help estimate which impact these changes in electrolytes have on the non-invasive glucose sensor.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age between 18 and 65 years

Exclusion Criteria:

* Uncontrolled hypertension (diastolic blood pressure > 100 mmHG and/or systolic blood pressure > 180 mmHg)
* Pregnancy or lactation period for female subjects
* Serious clinical signs of a liver disease, acute or chronic hepatitis, acute or chronic kidney disease, or ALAT > 2.5 times the upper level of normal values, or serum creatinine > 1.3 mg/dL (women)/1.5 mg/dL (men)
* Any serious acute illness (at the decision of the investigator), e.g. sepsis, gastric or duodenal ulcer, acute myocardial infarction, acute asthma attack
* Any other serious chronic illness (at the decision of the investigator), e.g. chronic obstructive pulmonary disease, any kind of cancer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2001-12; Primary Completion 2002-05 (Actual); Study Completion 2002-08 (Actual)

PRIMARY OUTCOMES:
plasma ion concentrations (sodium, potassium, chloride, calcium, magnesium) and osmolarity | blood samples every 10 min during baseline, plateau hyperglycemic and final euglycemic phase, every 5 min during increase and decrease of blood glucose

SECONDARY OUTCOMES:
blood glucose concentration | continuously during glucose clamp

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Kapitza, MD, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany